CLINICAL TRIAL: NCT04119999
Title: A Cardiosleep Research Program on Obstructive Sleep Apnea, Blood Pressure Control and Maladaptive Myocardial Remodeling
Acronym: CRESCENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: Ng Teng Fong General Hospital (Other); National University Hospital, Singapore (Other); National Heart Centre Singapore (Other)
Responsible Party: Principal Investigator, Chi-Hang Lee, Professor of Medicine, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Senior CSA
Record Dates: First submitted 2019-10-07; First posted 2019-10-09 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Hypertension,Essential; Obstructive Sleep Apnea
Keywords: sleep; remodeling; blood pressure; trial
MeSH Terms: conditions — Essential Hypertension; Sleep Apnea, Obstructive | interventions — Occlusal Splints; Continuous Positive Airway Pressure

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPAP (Active Comparator): Continuous Positive Airway Pressure
  Interventions: Device: Continuous Positive Airway Pressure
- MAD (Experimental): Mandibular Advancement Device
  Interventions: Device: Mandibular Advancement Device

INTERVENTIONS:
Device: Mandibular Advancement Device — Mandibular advancement device (MAD) has been a novel method in the management of snoring and OSA. For mild to moderate sleep apnea, MADs have been a boon. A guideline published by American Academy of Sleep Medicine stated that MAD was indicated as first-line therapy for mild OSA and a second-line therapy for moderate to severe OSA
  Arms: MAD
Device: Continuous Positive Airway Pressure — Continuous positive airway pressure (CPAP) is a form of positive airway pressure ventilator, which applies mild air pressure on a continuous basis to keep the airways continuously open in people with OSA
  Arms: CPAP

SUMMARY:
The objective of this proposal is to evaluate whether mandibular advancement device (MAD) is non-inferior to continuous positive airway pressure (CPAP) in the treatment of obstructive sleep apnea (OSA) and blood pressure reduction. OSA and hypertension are highly prevalent disorders with profound impacts on health. Apart from improving quality of-life, an effective OSA treatment could improve cardiovascular risk partly through blood pressure reduction, particularly in patients with high cardiovascular risk in whom blood pressure control is often suboptimal. Although CPAP is useful, the high non-acceptance and non-adherence preclude its widespread use.

East Asians have a restrictive craniofacial phenotype that predisposes them to OSA and the associated cardiovascular stress. CPAP, while considered the first-line therapy for OSA, has failed to improve cardiovascular outcomes in randomized trials till date because it is poorly tolerated. MADs are oral appliances that correct the restrictive craniofacial phenotype present in East Asians by protruding the lower jaw to reduce upper airway collapsibility. MADs are better tolerated than CPAP, and this may be an important determinant of the overall effectiveness in treating OSA, and thus ameliorating the downstream adverse health outcomes. We hypothesize that MADs are non-inferior to CPAP in treating OSA and reducing cardiovascular risk by blood pressure reduction in East Asians.

We will recruit East Asian subjects with hypertension and high cardiovascular risk for polysomnography. Patients diagnosed with OSA (n=220) will be randomized to MAD or CPAP groups in a 1:1 ratio for a treatment duration of 6 months. The primary endpoint is the 24-hour mean blood pressure as determined by ambulatory monitoring. The secondary endpoints include sleep-time systolic BP, target blood pressure, cardiovascular biomarkers, and myocardial remodeling. Association between OSA and silent paroxysmal atrial fibrillation will also be determined. If MADs are shown to be effective, the next step is to evaluate our novel device- drug-eluting MAD that the team is developing.

ELIGIBILITY:
Inclusion Criteria:

1. Age of at least 40 years
2. Chinese (based on the Identity Card or other Identity Document if the subject is a non-Singapore citizen or permanent resident)
3. Physician diagnosed essential hypertension, on at least 1 medication for BP control
4. High cardiovascular risk, as defined by one or more of the following: (a) diabetes mellitus, (b) stroke, (c) significant coronary artery disease (at least one stenosis of >50% diameter in at least one major epicardial artery), (d) chronic kidney disease, excluding polycystic kidney disease, with an estimated glomerular filtration rate of <60 ml/min/1.73m2, or (e) age of 75 years or older.

Exclusion Criteria:

1. Known OSA on treatment
2. Cheyne-Stokes breathing or predominantly central sleep apnea (>50%)
3. Known secondary hypertension: from renal (renal artery stenosis, chronic renal failure); endocrine (aldosterone excess, pheochromocytoma, cushing's syndrome, hyperthyroidism) or cardiac causes (aortic coarctation)
4. Contraindications to CMR: implantable devices, cerebral aneurysm clips, cochlear implants, renal impairment (GRF <30ml/min/1.73m2), claustrophobia and pregnant women
5. Contraindications to MAD: <6 to 10 teeth in each arch, inability to advance the mandible and open the jaw widely, pre-existing temporomandibular joint problems, severe bruxism
6. Limited life expectancy (< 1 year)
7. Hypertensive crisis, acute coronary syndromes or acute heart failure in the past 30 days
8. Known AF (not suitable for CMR and affects remodelling analysis)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
24-hour mean BP (24MBP) | 6 months
  Difference in 24-hour mean BP (24MBP) between the patients in the MAD and CPAP groups as determined by 24-hour ambulatory BP monitoring.

SECONDARY OUTCOMES:
24-hour systolic BP (24SBP) | 6 months and 12 months
  Difference in 24-hour systolic BP (24SBP) between the patients in the MAD and CPAP groups as determined by 24-hour ambulatory BP monitoring.
24-hour pulse pressure (24PP) | 6 months and 12 months
  Difference in 24-hour pulse pressure (24PP) between the patients in the MAD and CPAP groups as determined by 24-hour ambulatory BP monitoring.
Nocturnal dipping | 6 months and 12 months
  Difference in prevalence of nocturnal dipping between the patients in the MAD and CPAP groups as determined by 24-hour ambulatory BP monitoring.
Ectopic beat | 12 months
  Difference in prevalence of ectopic beats between the patients in the MAD and CPAP groups as determined by continuous ECG monitoring
Myocardial remodeling | 12 months
  Difference in LV and LA dimensions between the patients in the MAD and CPAP groups as determined by cardiac MRI
Epworth Sleepiness Scale (ESS) score | 6 months and 12 months
  Difference in change in ESS score between the MAD and CPAP groups
Sleep Apnea Quality of Life Index (SAQLI) | 6 months and 12 months
  Difference in change in SAQLI score between the MAD and CPAP groups
Functional Outcome of Sleep Questionnaire (FOSQ) | 6 months and 12 months
  Difference in change in SAQLI score between the MAD and CPAP groups
36-Item Short Form Health Survey (SF-36) | 6 months and 12 months
  Difference in change in SF-36 score between the MAD and CPAP groups
EuroQol 5Q (EQ5D) | 6 months and 12 months
  Difference in change in EQ5D score between the MAD and CPAP groups
Daytime systolic BP | 6 months and 12 months
  Difference in change in daytime systolic BP between the patients in the MAD and CPAP
Nighttime systolic BP | 6 months and 12 months
  Difference in change in nighttime systolic BP between the patients in the MAD and CPAP
Percentage of patient with 24-hour systolic BP<130 mmHg | 6 months and 12 months
  Difference in percentage of patients with 24-hour systolic BP<130 mmHg in the MAD and CPAP groups
Percentage of patient with 24-hour systolic BP<120 mmHg | 6 months and 12 months
  Difference in percentage of patients with 24-hour systolic BP<120 mmHg in the MAD and CPAP groups
NT-proBNP | 6 months and 12 months
  Change in the plasma level of NT-proBNP from baseline to 6-month follow-up
High sensitivity troponin | 6 months and 12 months
  Change in the plasma level of high sensitivity troponin from baseline to 6-month follow-up
High sensitive C-reactive protein | 6 months and 12 months
  Change in the plasma level of high sensitive C-reactive protein from baseline to 6-month follow-up

OTHER OUTCOMES:
Subgroup analysis | 6 months and 12 months
  Prespecified subgroups include - Age, Gender, BMI, wrist circumference, AHI, ODI, ESS, DM, IHD, number of HT medicine, Device adherence

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Hang Lee, MD, Principal Investigator — National University of Singapore
Locations (1):
- NUHS Cardiosleep research laboratory, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided
The individual participant data generated by the CRESCENT trial will be made available as soon as possible upon reasonable request, wherever legally and ethically possible.

REFERENCES:
- [Derived] Colpani JT, Ou YH, Kosasih AM, Lee FKF, Chan SP, Tan HH, Wong RCW, Chin CW, Cistulli PA, Lee CH. Mandibular Advancement Device versus CPAP in Severe Obstructive Sleep Apnea. J Dent Res. 2026 Jan;105(1):112-119. doi: 10.1177/00220345251361796. Epub 2025 Sep 1. PMID 40888163
- [Derived] Colpani JT, Ou YH, Thakumar AV, Cheong CS, Loke W, Sia CH, Teo YH, Chan SP, Chin CW, Kojodjojo P, Chan MY, Cistulli PA, Luo N, Lee CH. Patient-reported quality of life outcomes with mandibular advancement versus continuous positive airway pressure: insights from the CRESCENT trial. Sleep. 2025 Nov 10;48(11):zsaf022. doi: 10.1093/sleep/zsaf022. PMID 39887015
- [Derived] Ou YH, Colpani JT, Cheong CS, Loke W, Thant AT, Shih EC, Lee F, Chan SP, Sia CH, Koo CY, Wong S, Chua A, Khoo CM, Kong W, Chin CW, Kojodjojo P, Wong PE, Chan MY, Richards AM, Cistulli PA, Lee CH. Mandibular Advancement vs CPAP for Blood Pressure Reduction in Patients With Obstructive Sleep Apnea. J Am Coll Cardiol. 2024 May 7;83(18):1760-1772. doi: 10.1016/j.jacc.2024.03.359. Epub 2024 Apr 6. PMID 38588926
- [Derived] Ou YH, Colpani JT, Chan SP, Loke W, Cheong CS, Kong W, Chin CW, Kojodjojo P, Wong P, Cistulli P, Lee CH. Mandibular advancement device versus CPAP in lowering 24-hour blood pressure in patients with obstructive sleep apnoea and hypertension: the CRESCENT trial protocol. BMJ Open. 2023 May 31;13(5):e072853. doi: 10.1136/bmjopen-2023-072853. PMID 37258080